CLINICAL TRIAL: NCT05281783
Title: Efficacy and Response Predictors of Percutaneous Radiofrequency Ablation for Treatment of Intermediate Stage Hepatocellular Carcinoma: A Controlled Clinical Trial
Brief Title: RFA for Treatment of Intermediate Stage HCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Collaborators: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Manar Ahmed Kamal, Principal Investigator, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMBSUREC/10102021/Eid
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Percutaneous Radiofrequency Ablation; Intermediate Stage; Hepatocellular Carcinoma; Clinical Trial
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: Single-center, prospective non-randomized, controlled clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Percutaneous Radiofrequency Ablation (Experimental): We aim to evaluate the percutaneous radiofrequency ablation (RFA) efficacy as monotherapy in intermediate versus early-stage hepatocellular carcinoma (HCC).
  Interventions: Device: percutaneous radiofrequency ablation (RFA)

INTERVENTIONS:
Device: percutaneous radiofrequency ablation (RFA) — We aim to evaluate the percutaneous radiofrequency ablation (RFA) efficacy as monotherapy in intermediate versus early-stage hepatocellular carcinoma (HCC).

SUMMARY:
In Egypt, chronic hepatitis C virus (HCV) is the most prevalent cause of hepatoma. The study aims to evaluate the percutaneous radiofrequency ablation (RFA) efficacy as monotherapy in intermediate versus early-stage hepatocellular carcinoma (HCC). The present study was a single-center, prospective non-randomized, controlled clinical trial in the Interventional Ultrasonography Unit, Tropical Medicine Department, Beni-Suef University Hospitals, between October 2018 and August 2021. Abdominal ultrasonography and triphasic computerized tomography (CT) abdomen were used to diagnose HCC. The abdominal ultrasonography and a dynamic CT scan were performed six weeks following the ablation to assess treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients were early and intermediate-stage HCC (BCLC stage A and B).
* Patients accepted to be treated by percutaneous radiofrequency ablation in the Interventional Ultrasonography Unit.
* Patients with early-stage-HCC should have up to 3 tumors, all smaller than 3 cm with a Child-Pugh A score.
* Patients with intermediate-stages-HCC should have multinodular HCC (>3 nodules <3 cm) or single focal lesion more than 3 cm, with Child-Pugh Score A or B liver cirrhosis, international normalized ratio (INR) less than 1.7, and platelet count more than 50,000/cm.

Exclusion Criteria:

* Patients with HCC with and vascular spread (portal vein thrombosis), lymph node metastasis or distant metastasis, subcapsular lesions, or lesions with close vicinity to the gall bladder, bowel, or portal vein.
* Patients with clinically decompensated liver disease (Child-Pugh Score C liver cirrhosis).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
The efficacy | six weeks after the date of the last ablation
  By evaluating the HCC biomarkers as serum AFP and VEGF

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety] | six weeks after the date of the last ablation
  By accounting for the number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ragaey A Eid, Principal Investigator — ragaeyahmad@med.bsu.edu.eg
Locations (1):
- Interventional Ultrasonography Unit, Tropical Medicine Department, Beni-Suef University Hospitals, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: Undecided